CLINICAL TRIAL: NCT01781637
Title: Phase 2 Study of Omalizumab in Oral Peanut Desensitization
Brief Title: Peanut Reactivity Reduced by Oral Tolerance in an Anti-IgE Clinical Trial
Acronym: PRROTECT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Stanford University (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Lynda Schneider, Professor, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Peanut 002
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Peanut Allergy; Food Allergy
Keywords: Xolair; omalizumab; peanut; oral desensitization
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- omalizumab group (Experimental): Patients will receive omalizumab.
  Interventions: Drug: Omalizumab
- placebo (Placebo Comparator): Patients will receive placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Omalizumab — subcutaneous injection
  Other Names: Xolair
  Arms: omalizumab group
Drug: placebo — subcutaneous injection
  Arms: placebo

SUMMARY:
The investigators will perform a double blind, placebo controlled clinical trial with Xolair (omalizumab) at four centers to safely and rapidly desensitize patients with severe peanut allergy. The investigators will determine if pretreatment with anti-IgE mAb (Xolair/omalizumab) can greatly reduce allergic reactions and allow for faster and safer desensitization.

DETAILED DESCRIPTION:
36 subjects will receive Xolair, and 8 subjects will receive placebo. The study will occur at 4 sites: Boston Children's Hospital, Children's Hospital of Philadelphia, Stanford University and Lurie Children's Hospital.

Patients will be pre-treated with Xolair or placebo before rapid oral peanut desensitization. Patients will continue to receive Xolair during the 8 subsequent weeks of desensitization, receiving their final dose of Xolair one week after reaching the highest tolerated dose of peanut.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe peanut allergy-sensitive subjects between the ages of 7 to 25 years old.
* Sensitivity to peanut allergen will be documented by a positive skin prick test result (6 mm diameter wheal or greater)
* ImmunoCAP IgE level to peanut > 10 kU/L.
* Sensitivity to peanut allergen based on a double-blind placebo-controlled oral food challenge (DBPCFC) at maximum of cumulative 175 mg of peanut protein dose.

Exclusion Criteria:

* Subjects with a total IgE at screening of < 50 kU/L > 2,000 kU/L.
* Positive reaction to the placebo on DBPCFC.
* Previous reaction to omalizumab.
* Subjects having a history of severe anaphylaxis to peanut requiring intubation or admission to an ICU, frequent allergic or non-allergic urticaria, or history consistent with poorly controlled persistent asthma, or gastrointestinal or gastroesophageal disease.

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda C Schneider, MD, Principal Investigator — Boston Children's Hospital; Andrew MacGinnitie, MD, PhD, Study Chair — Children' Hospital Boston; Kari Nadeau, MD, PhD, Study Chair — Stanford University; Jonathan Spergel, MD, PhD, Study Chair — Children's Hospital of Philadelphia; Jacqueline Pongracic, MD, Study Chair — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Lurie Children's Hospital, Chicago, Illinois
  - Division of Immunology, Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen G, Shrock EL, Li MZ, Spergel JM, Nadeau KC, Pongracic JA, Umetsu DT, Rachid R, MacGinnitie AJ, Phipatanakul W, Schneider L, Oettgen HC, Elledge SJ. High-resolution epitope mapping by AllerScan reveals relationships between IgE and IgG repertoires during peanut oral immunotherapy. Cell Rep Med. 2021 Oct 19;2(10):100410. doi: 10.1016/j.xcrm.2021.100410. eCollection 2021 Oct 19. PMID 34755130

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab Group | Placebo
Started | 28 | 8
Completed | 24 | 2
Not Completed | 4 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 2 | 6
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab Group | Placebo | Total
Number analyzed (Participants) | 29 | 8 | 37
Age, Continuous [Median (Full Range); unit: years] | 10 [7 to 19] | 10 [6 to 17] | 10 [6 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 18 | 4 | 22
Baseline population [Count of Participants; unit: Participants] — Population: One subject declined treatment after being randomized but before beginning treatment
  Participants | 29 | 8 | 37

OUTCOME MEASURES:

1. Primary Outcome: Tolerance of 2000 mg 6 Weeks After Last Dose of Omalizumab/Placebo
Time Frame: 6 weeks after last dose of omalizumab/placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab Group | Placebo
Number analyzed (Participants) | 29 | 8
Participants | 23 | 1

2. Secondary Outcome: Pass 4000 mg OFC 12 Weeks After Last Dose of Omalizumab/Placebo
Time Frame: 12 weeks after last dose of omalizumab/placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Omalizumab Group | Placebo
Number analyzed (Participants) | 29 | 8
Participants | 20 | 1

ADVERSE EVENTS:
Arm/Group | Omalizumab Group | Placebo
Serious Adverse Events (participants affected / at risk) | 4/28 | 3/8
Other Adverse Events (participants affected / at risk) | 28/28 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab Group (N=28) | Placebo (N=8)
Anaphylaxis (Immune system disorders) | 3 (3) | 3 (3)
Psychiatric (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab Group (N=28) | Placebo (N=8)
Abdominal Pain (Gastrointestinal disorders) | 10 | 5
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Anaphylaxis (Immune system disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 0
Fever (General disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 11 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No